CLINICAL TRIAL: NCT01967082
Title: APPSPIRE: Expanding the Reach of an Innovative Tobacco Control Program for Youth
Brief Title: APPSPIRE App in Preventing Students From Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-0369; NCI-2018-03054 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0369 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); R41DA035012 (NIH)
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Cigarette Smoker; Current Every Day Smoker; Student
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (focus group, APPSPIRE app, survey) (Experimental): Participants attend an audio-taped focus group over 1 hour and are given the APPSPIRE app. After 1 and 4 months of using the app, participants complete a telephone survey over 1 hour to discuss how they liked the app and its usefulness.
  Interventions: Behavioral: APPSPIRE; Behavioral: Focus Group; Other: Survey Administration

INTERVENTIONS:
Behavioral: APPSPIRE — Given APPSPIRE app
  Other Names: APPSPIRE Smartphone Application; APPSPIRE Smartphone App; APPSPIRE App; APPSPIRE Application
Behavioral: Focus Group — Attend focus group
Other: Survey Administration — Complete survey

SUMMARY:
This trial studies how well APPSPIRE, a smartphone app, works in preventing students from smoking. Technology-driven intervention programs, such as the APPSPIRE app, have the potential to increase access to health behavior treatments and therapies, such as tobacco cessation support, and provide effective prevention messaging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop a prototype of the APPSPIRE (phone application [app] of a smoking prevention interactive experience).

II. At post assessment, students enrolled in the study will qualitatively provide information about the usability and usefulness for the prevention and cessation sites.

III. Investigate frequency of use of and exposure to APPSPIRE modules via an objective measure of general use.

IV. Investigate how feasible the program will be. V. Obtain a maintained use of APPSPIRE with high completeness and extent of completion.

VI. Evaluate change in stage of change from baseline to about 1 and 4-month follow-ups among participants.

OUTLINE:

Participants attend an audio-taped focus group over 1 hour and are given the APPSPIRE app. After 1 and 4 months of using the app, participants complete a telephone survey over 1 hour to discuss how they liked the app and its usefulness.

ELIGIBILITY:
Inclusion Criteria:

* Student at Houston Community College (HCC)
* Speak and read English
* Own an iPhone
* Be enrolled in at least one class at HCC
* Provide current contact information
* Smoke 1 or more cigarettes a day (cessation group)
* Have access to the internet (cessation and prevention/advocacy groups)
* Evidence of smoking susceptibility as defined by the Smoking Susceptibility Scale

Exclusion Criteria:

* Does not plan to continue as a student at their campus sometime during the year of the study (cessation and prevention/advocacy groups)
* Current tobacco use (prevention/advocacy group)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Frequency of APPSPIRE application (app) use | Up to 4 months
  Will be measured in minutes per day and with descriptive statistics. Will measure using mean, median and standard deviation for continuous variables.
The Feasibility of the tobacco control program. | Up to 4 months
  Feasibly will be measured by multiplying the variable of two concepts: ease of use and ability to fit the program into routine schedules.
The Completeness with the Percentages of Participants surveyed. | Up to 4 months
  Completeness will be measured as the percentage of participants who continue to use AppSPIRE until the 4 month follow up survey.
The extent of completion for the modules AppSPIRE. | Up to 4 months
  The extent of completion includes the various modules of AppSPIRE. High extent of completion is obtained if 75% of the participants have completed all modules of AppSPIRE.
The Stages of the Change Scale | Baseline up to 4 months
  A validated measure, The Stages of Change Scale, will be used to clarify smokers into 3 categories: pre-contemplation, contemplation and preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Prokhorov, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Houston Community College, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org